CLINICAL TRIAL: NCT05752214
Title: Observational Study on Quality of Life in Visually Impaired Patients Through the Questionnaire VA LV VFQ in Italy
Brief Title: Quality of Life in Italian Visually Impaired Patients
Acronym: SOPIITA
Status: Recruiting | Type: Observational
Sponsor: Amore Filippo (Other)
Responsible Party: Sponsor-Investigator, Amore Filippo, Medical Doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Organization: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Other Study IDs: 3904
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Visual Impairment
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group A
  Interventions: Other: WEB Register

INTERVENTIONS:
Other: WEB Register — Observational, non-profit, multicentre longitudinal study on the assessment of quality of life and its association with demographic variables and visual function of visually impaired patients attending the visual rehabilitation service.

SUMMARY:
Clinical register of visual rehabilitation activity and observational study on the validation of the VA LV VFQ questionnaire in the Italian context

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years or older, suffering from any visual pathology, who are admitted to specialised visual rehabilitation centres for visual rehabilitation.
* Ability to understand and sign the informed consent for participation in the study.

Exclusion Criteria:

* Less than 18 years of age.
* Cognitive impairment that, in the opinion of the investigator, limits understanding of the informed consent or the questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Visually impaired subjects
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
VA-LV-VFQ-48 questionnaire score | 10 years
  Clinical register of visual rehabilitation activity and observational study on the validation of the VA LV VFQ questionnaire in the Italian context

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No